CLINICAL TRIAL: NCT02154958
Title: Role of Follicular Output Rate in the Prediction of in Vitro Fertilization and Intracytoplasmic Sperm Injection Outcome in Women With Unexplained Infertility
Brief Title: Role of Follicular Output Rate in the Prediction of in Vitro Fertilization and Intracytoplasmic Sperm Injection in Women With Unexplained Infertility
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, AbdelGany Hassan, Lecturer, Cairo University
Other Study IDs: Sub 1
Record Dates: First submitted 2014-05-28; First posted 2014-06-04 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Subfertility; Assisted Reproduction
Keywords: Follicular output rate; IVF; ICSI
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Unexplained infertility

SUMMARY:
300 women with unexplained infertility who are already decided to be treated with ICSI will be recruited from Cairo university hospitals and Dar Al-Teb subfertility centre.

On the second day of menstruation serum FSH, LH, Prolactin and Oestradiol will be assessed and the antral follicular count (AFC) will be assessed using a vaginal ultrasound scan. AFC will be defined as the number of follicles measuring 3-10mm.

All patients will have standard pituitary down-regulation followed by (Human menopausal gonadotrophin (HMG) stimulation until the day of (Human chorionic gonadotrophin (HCG) administration. On the day of HCG administration, ovarian ultrasound scan will be performed using a transvaginal probe and the Preovulatory follicle count (PC) will be assessed, (PFC) is defined as number of follicles measuring≥16mm. FORT will be calculated as: (PFC) * 100/AFC.

DETAILED DESCRIPTION:
Our study is observational, we are observing data from routine measurements during IVF/ICSI. Our study does not assess IVF/ICSI as an intervention, we are evaluating the role of FORT which is calculated by observing routine measurements during the IVF/ICSI procedure.

300 women with unexplained infertility who are already decided to be treated with ICSI will be recruited from Cairo university hospitals and Dar Al-Teb subfertility centre.

All women fulfilling the inclusion criteria will be invited to participate in the study. A written informed consent will be taken and only women signing the consent will be included in the study. Patients included in the study will be subjected to full history taking and clinical examination including general, abdominal and gynecological examination. This will be followed by a vaginal ultrasound scan to assess uterus, ovaries and any pelvic masses.

All women will go through the usual IVF/ICSI procedure explained below, our aim is to observe the antral follicle count, the pre-ovulatory count and calculate the FORT then correlating this with pregnancy.

On the second day of menstruation serum FSH, LH, Prolactin and Oestradiol will be assessed and the antral follicular count (AFC) will be assessed using a vaginal ultrasound scan. AFC will be defined as the number of follicles measuring 3-10mm.

All patients will have standard pituitary down-regulation protocol with GnRHa (Triptorelin 0.1mg, Decapeptyl® Ferring, Germany) day 7 after ovulation of previous cycle or on day 21 of the oral contraceptive cycles. GnRHa will be continued for 2 weeks. Human menopausal gonadotrophin(HMG) (Merional ®IBSA) 150-300 IU/day will be administered until the day of HCG administration.

On the day of HCG administration, ovarian ultrasound scan will be performed using a transvaginal probe and the Preovulatory follicle count (PC) will be assessed, (PFC) is defined as number of follicles measuring≥16mm. FORT will be calculated as: (PFC) * 100/AFC.

FORT values will be classified into 3 categories: low, medium and high the 3 groups will be compared regarding the clinical pregnancy rate, number of retrieved oocytes, number and quality of embryos The procedure will be cancelled if less than 3 follicles 16-20 mm in size are present 12 days after starting FSH despite doses reaching 450 IU. The cycle will be also cancelled if there is risk of ovarian hyperstimulation like massive ovarian enlargement or serum estradiol exceeds 3000pg/L Transvaginal oocyte retrieval will be performed 34-36 h after the administration of HCG. Oocytes will be fertilized either via IVF or ICSI based on the couple's history. Fertilization will be assessed 16-18 h after IVF or ICSI. Embryo transfers will be performed 3 days after oocyte retrieval. No more than three embryos per patient will be transferred; vaginal tablets containing progesterone (Prontogest® IBSA) administered 400 mg/day as luteal support from the day of the oocyte retrieval. Clinical pregnancy will be defined as Visualization of an intrauterine gestational sac 5 weeks after embryo transfer.

ELIGIBILITY:
Inclusion Criteria:

* Unexplained infertility
* Both ovaries are present
* Day 2 FSH <10 mIU/L
* Day 2 Estradiol <80 pg/L

Exclusion Criteria:

* Known other cause of subfertility
* Expected poor responders according to Bologna criteria (9)
* Abnormalities affecting the uterine cavity
* Uncontrolled diabetes
* Allergy to gonadotrophins
* Cancelled cycles during the study

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: 300 women with unexplained infertility who are already decided to be treated with ICSI will be recruited
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2014-05; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy | 5 weeks after embryo transfer
  FORT values will be classified into 3 categories: low, medium and high. The proportion of women achieving a clinical pregnancy will be compared among the 3 groups. Clinical pregnancy will be defined as the presence of an intra-uterine gestational sac detected by ultrasound scanning.

SECONDARY OUTCOMES:
Retrieved oocytes | 1 hour after ovum pick up
  FORT values will be classified into 3 categories: low, medium and high. The number of retrieved oocytes will be compared among the 3 groups.
Number of embryos | 3 days after ovum pick up
  FORT values will be classified into 3 categories: low, medium and high. The number of embryos will be compared among the 3 groups
Quality of embryos | 3 days after ovum pick up
  FORT values will be classified into 3 categories: low, medium and high. Embryo quality will be categorised fro 1-4 according to the symmetry of cells, cell fragmentation and the number of cells. The 3 groups will be compared regarding the quality of embryos

CONTACTS AND LOCATIONS:
Overall Officials: AbdelGany MA Hassan, MRCOG, MD, Principal Investigator — Cairo University
Locations (2):
- Egypt (2):
  - Cairo University Hospitals, Cairo
  - Dar AlTeb subfertility centre, Giza

REFERENCES:
- [Background] Brandes M, Hamilton CJ, van der Steen JO, de Bruin JP, Bots RS, Nelen WL, Kremer JA. Unexplained infertility: overall ongoing pregnancy rate and mode of conception. Hum Reprod. 2011 Feb;26(2):360-8. doi: 10.1093/humrep/deq349. Epub 2010 Dec 16. PMID 21163857
- [Background] Zhang N, Hao CF, Zhuang LL, Liu XY, Gu HF, Liu S, Chen ZJ. Prediction of IVF/ICSI outcome based on the follicular output rate. Reprod Biomed Online. 2013 Aug;27(2):147-53. doi: 10.1016/j.rbmo.2013.04.012. Epub 2013 May 4. PMID 23768619
- [Background] de Carvalho BR, Rosa e Silva AC, Rosa e Silva JC, dos Reis RM, Ferriani RA, Silva de Sa MF. Ovarian reserve evaluation: state of the art. J Assist Reprod Genet. 2008 Jul;25(7):311-22. doi: 10.1007/s10815-008-9241-2. Epub 2008 Aug 5. PMID 18679790
- [Background] Broer SL, Mol BW, Hendriks D, Broekmans FJ. The role of antimullerian hormone in prediction of outcome after IVF: comparison with the antral follicle count. Fertil Steril. 2009 Mar;91(3):705-14. doi: 10.1016/j.fertnstert.2007.12.013. Epub 2008 Mar 5. PMID 18321493
- [Background] Melo MA, Garrido N, Alvarez C, Bellver J, Meseguer M, Pellicer A, Remohi J. Antral follicle count (AFC) can be used in the prediction of ovarian response but cannot predict the oocyte/embryo quality or the in vitro fertilization outcome in an egg donation program. Fertil Steril. 2009 Jan;91(1):148-56. doi: 10.1016/j.fertnstert.2007.11.042. Epub 2008 May 2. PMID 18455166
- [Background] Genro VK, Grynberg M, Scheffer JB, Roux I, Frydman R, Fanchin R. Serum anti-Mullerian hormone levels are negatively related to Follicular Output RaTe (FORT) in normo-cycling women undergoing controlled ovarian hyperstimulation. Hum Reprod. 2011 Mar;26(3):671-7. doi: 10.1093/humrep/deq361. Epub 2010 Dec 21. PMID 21177311